CLINICAL TRIAL: NCT03889483
Title: Neurophysiological Measurements in the Pediatric Concussion Population: An Initial Assessment Using the NeuroCatch™ Platform
Brief Title: Neurophysiological Measurements Using the NeuroCatch™ Platform in Pediatric Concussion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Michael Esser (Other)
Collaborators: NeuroCatch Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dr. Michael Esser, Principal Investigator, Alberta Children's Hospital
Organization: Alberta Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACH-NCI-001
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Children, Only; Traumatic Brain Injury; Concussion, Mild; Pediatric ALL
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Participants will be divided into the following cohorts:
  Cohort 1: 30 participants with persistent mTBI symptoms (duration greater than 6 weeks), as determined by the Investigator; Cohort 2: 30 participants who recovered quickly from mTBI (i.e., within approximately six weeks based on symptomatology), as determined by the Investigator; Cohort 3: 15 participants who have had multiple mTBIs (2 or more medically verified concussions over the last year); and Cohort 4: 30 participants who have never had a concussion. Participants in Cohorts 1-3 will be recruited 6-16 weeks post injury date.
  After study enrollment, all participants undergo two NeuroCatch Platform assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeuroCatch™ Platform Assessment (Other): All participants will undergo two NeuroCatch™ Platform Assessments.
  Interventions: Device: NeuroCatch™ Platform

INTERVENTIONS:
Device: NeuroCatch™ Platform — The NeuroCatch™ Platform consists of software and hardware that captures brain health information. The platform intends to provide a quick, portable and easy to use solution for the acquisition, display, analysis, storage, reporting and management of electroencephalograph (EEG) and event-related potential (ERP) information.

SUMMARY:
EEG signals have been collected and studied since the early 1990's as a way of assessing brain function at a gross level. As early as the 1930's a derivative of the raw EEG signal - event-related potentials (ERPs) - have been computed. The current research is primarily focused on three ERP components: the N100, P300 and N400. Each of the three ERPs have been studied in the academic laboratory for multiple decades. Through this research, a strong understanding has been developed regarding what can affect these components (e.g. task set, emotional state, etc.). However, these signals within various pediatric populations (e.g., those with persistent mTBI symptoms or multiple concussions) are not well characterized.

Being able to safely and effectively employ the NeuroCatch™ Platform in a post-concussive pediatric cohort could provide researchers with the potential to elucidate the persistence of objective measures of impairment, patterns of recovery, and chronicity of problems due to mTBI in children. Secondly, understanding the degree to which these neurophysiological components fluctuate over time is crucial to the understanding of brain functioning. However, for this type of technology to be useful in quantifying brain health in this population,the degree to which a post-concussive pediatric brain naturally fluctuates in its processing capability must be quantified. NeuroCatch™ Platform has the ability to measure changes in several domains of brain function. These cognitive processes are foundational blocks for some of the highest cognitive processes: information integration and executive functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Male, female, or intersex
2. 8-18 years old inclusively
3. Must meet all criteria in one of the following cohorts:

   1. Cohort 1: Has persistent mTBI symptoms 6-16 weeks post-injury, as determined by the Investigator;
   2. Cohort 2: Recovered quickly (within approximately six weeks) from mTBI, as determined by the Investigator 6-16 weeks post-injury;
   3. Cohort 3: Has had multiple mTBIs (2 or more medically verified concussions over the last year) with the most recent injury having occurred 6-16 weeks prior to study enrollment;
   4. Cohort 4: Has never had a concussion.

Exclusion Criteria:

1. Previous neurological illnesses (e.g., epilepsy or seizure disorders) including moderate to severe learning difficulties, as determined by the Investigator
2. Clinically documented hearing issues (e.g., tinnitus, in-ear hearing problems, punctured ear drum)
3. In-ear hearing aid or cochlear implant, hearing devices
4. Implanted pacemaker
5. Metal or plastic implants in skull
6. Allergy to rubbing alcohol or EEG gel
7. Previous participation in one or more studies using the NeuroCatchTM Platform
8. Unhealthy scalp (apparent open wounds and/or bruised or weakened skin)
9. Using other investigational drugs or devices while enrolled in this study
10. Not fluent in the English language
11. If female and of child-bearing potential: suspected or planning to become pregnant, currently pregnant, or breast-feeding

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 105 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Tracking and comparison of neurophysiological changes (ERP response size) to persistence of mTBI symptoms | 1 day
  Response size will be measured as amplitude in microvolts. Persistence of mTBI symptoms will be defined by cohort.
Tracking and comparison of neurophysiological changes (ERP response timing) to persistence of mTBI symptoms | 1 day
  Response timing will be measured as latency in milliseconds. Persistence of mTBI symptoms will be defined by cohort.

SECONDARY OUTCOMES:
Number of adverse events and adverse device effects | 1 day
  Assessing the safety and performance of the NeuroCatchTM Platform in four pediatric cohorts.
Collection of ERP response size (amplitude in microvolts) and response timing (latency in milliseconds) | 1 day
  Quantifying the natural variability in selected ERPs (N100, P300, N400) acquired using the NeuroCatchTM Platform in one study session.

OTHER OUTCOMES:
Explore trends between select additional measures of impairment and ERPs across four pediatric cohorts. | 1 day
  Additional measures of impairment may include cognitive assessments, blood work and DNA analysis, brain imaging (MRI) and levels of carbon dioxide in the breath.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Esser, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Department of Paediatrics, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided